CLINICAL TRIAL: NCT06469736
Title: Standard of Care Ureterorenoscopy With Lithotripsy Versus in Combination With the Hydrogel Method for Kidney Stone Removal: An Open, Randomized, Monocentric Study
Brief Title: Comparison Between Ureterorenoscopy With Lithotripsy Alone Versus Combination With Hydrogel for Kidney Stone Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Thomas Amiel, Medical Doctor, Technical University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-395-S-KK
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Nephrolithiasis; Lithotripsy, Laser; Ureteroscopy
Keywords: Hydrogel; MediNiK; Hydrogel methode; Stone Free Rate; Zero Residual Fragments; URS; Dusting; Stone free; Thulium; Kidneystones
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Ureterorenoscopy (Sham Comparator): Arm A) Standard procedure ( URS) for the removal of kidney stones using URS
  Interventions: Procedure: Standard of Care Ureterorenoscopy
- Standard of Care Ureterorenoscopy with MediNik (Active Comparator): Arm B) Standard procedure (URS) for the removal of kidney stones using URS in combination with the mediNiK®
  Interventions: Procedure: Standard of Care Ureterorenoscopy with MediNiK

INTERVENTIONS:
Procedure: Standard of Care Ureterorenoscopy — The patient provides written informed consent and is positioned in the supine position. After disinfection, sterile draping, and single-shot antibiotic administration a rigid cystoscopy is performed. Intubation of the ostium with a hydrophilic guidewire and placed into the renal pelvis under fluoroscopic control. After a semirigid URS, a working sheath is placed up to the Kidney. A flexible URS with lithotripsy with a Thulium lase is then performed to dust the stones. The fragments are retrieved for analysis. Finally, a double-J or mono-J stent and a transurethral catheter are placed.
  Arms: Standard of Care Ureterorenoscopy
Procedure: Standard of Care Ureterorenoscopy with MediNiK — The patient provides written informed consent and is positioned in the supine position. After disinfection, sterile draping, and single-shot antibiotic administration a rigid cystoscopy is performed. Intubation of the ostium with a hydrophilic guidewire and placed into the renal pelvis under fluoroscopic control. After a semirigid URS, a working sheath is placed up to the Kidney. A flexible URS with lithotripsy with a Thulium lase is then performed to dust the stones. The fragments are retrieved for analysis. Application of MediNiK to embbed the residual stones in the hydrogel and extract it with a basket. Finally, a double-J or mono-J stent and a transurethral catheter are placed.
  Arms: Standard of Care Ureterorenoscopy with MediNik

SUMMARY:
The incidence of kidney stones (urolithiasis) has surged in both developing and developed countries, affecting approximately 15% of the global population. From 2010 to 2019, diagnoses of kidney and ureteral stones rose by 8% in Germany, 26% in France, and 15% in England. Correspondingly, the number of surgical stone removal procedures increased by 3%, 38%, and 18%, respectively. Common treatments include extracorporeal shock wave lithotripsy (ESWL), ureterorenoscopy (URS) with lithotripsy, and percutaneous nephrolithotomy (PCNL).

URS, depending on stone size, has become a preferred method due to advancements in intraoperative imaging and laser technology. Despite these improvements, small fragments often remain post-intervention, leading to recurrent stones. Complete removal of all fragments is crucial to significantly reduce recurrence rates. Current literature suggests a high recurrence rate with residual fragments, impacting healthcare costs and patient quality of life.

A key objective in endourological research is optimizing the stone clearance rate. Techniques like coagulum lithotomy and the autologous blood clot technique have been developed to enhance residual stone removal after laser fragmentation. These methods benefit selected patients but are not widely adopted due to complications such as reduced intraoperative visibility and long coagulum formation times.

Recently, a two-component hydrogel system called mediNiK® (Purenum GmbH, Germany) was developed. This biocompatible gel can be applied through an endoscope after stone fragmentation and large fragment retrieval to embed smaller fragments and dust, forming a removable conglomerate. MediNiK® has demonstrated effectiveness in embedding and removing stone residues and is already in clinical use in Europe, showing potential for optimizing stone removal.

A multicenter study has assessed the safety and tolerability of mediNiK® in standard URS (Open, randomized, multicentre study to evaluate the safety, tolerability, and performance of mediNiK® compared to standard treatment in kidney stone removal - DRKS00030532). Results indicate the gel is safe and tolerable. However, further data from larger cohorts and comparisons with conventional URS are necessary before widespread adoption of mediNiK®.

DETAILED DESCRIPTION:
The incidence of kidney stones (urolithiasis) has increased in both developing and developed countries, affecting around 15% of the world's population (1). Between 2010 and 2019, the diagnosis of kidney and ureteral stones in Germany, France and England increased by 8%, 26% and 15% respectively, while the number of surgical procedures to remove stones increased by 3%, 38% and 18% respectively (2). Common surgical treatments for kidney stones include extracorporeal shock wave lithotripsy (ESWL), ureterorenoscopy (URS) with lithotripsy and percutaneous nephrolithotomy (PCNL).

Depending on the size of the stone, URS has sometimes established itself as the method of choice, not least thanks to improved intraoperative imaging and the further development of laser technology. Despite these innovations, small fragments can remain in the kidney post-intervention, which in turn can lead to new stone formation (recurrent stones). From a medical point of view, complete removal of all fragments is essential in order to significantly reduce the recurrence rate of affected patients. According to the current literature, the recurrence rate in the sense of so-called secondary stone formation is estimated to be high in the case of residual fragments (3), associated with associated costs for the healthcare system and restrictions in the quality of life of the affected patients.

A major goal of endourological research in this area is therefore to optimize the stone clearance rate. Procedures such as coagulum lithotomy or the "autologous blood coagel technique" have been developed to improve the removal of residual stones after laser-guided fragmentation. Selected patients can benefit from these techniques, but their widespread use is limited, particularly due to the often associated deterioration in intraoperative visibility and the long waiting times until coagulum formation (4). For this reason, a two-component hydrogel system called mediNiK® (Purenum GmbH, Germany) was recently developed. This gel, consisting of two biocompatible components, can be applied via the inserted endoscope in a controlled manner and under visualization after completion of stone fragmentation and retrieval of large fragments in order to embed smaller stone fragments and dust. The resulting conglomerate can then be removed using conventional grasping forceps (5).

The hydrogel method with mediNik® has proven to be effective in embedding and removing stone residues (6). The system is already being used clinically in Europe and shows great potential for optimizing stone removal. A safety assessment in a multicenter study has already shown that the use of the gel is safe and tolerable in the context of standard URS. (Open, randomized, multicentre study to evaluate the safety, tolerability and performance of mediNiK® compared to standard treatment in the removal of kidney stones - DRKS00030532 - https://drks.de/search/de/trial/DRKS00030532.) However, before mediNik® can be used across the board, further data in a larger cohort and, in particular, a comparison with conventional URS are required.

The primary objective of this study is to compare the standard URS for the treatment of kidney stones without and with mediNik® with regard to the postoperative stone clearance rate. Further secondary endpoints are described in chapter 4. The results should provide the central basis for optimizing stone therapy at European centers and thereby improving medical care while optimizing costs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years
* Evidence of nephrolithiasis on presentation of a preoperative computer tomography (CT) scan not older than 6 months
* Minimum size of the kidney stones defined as >10mm in the longest axis in the preoperative CT.
* Ability to read, write and speak German
* Women of childbearing age must have a negative serum pregnancy test at the start of the study.
* Submission of a personally signed and dated informed consent form stating that the subject has been informed of all relevant aspects of the study prior to any trial-related activity and that all information has been understood

Exclusion Criteria:

* Participation in another clinical trial for kidney stone removal in the last 6 months
* Subjects with gastrointestinal cancer who have not been in remission for at least 2 years
* Subjects with a single kidney, horseshoe kidney or other anatomical abnormalities that may increase the risk of surgery for the subject
* Subjects with untreated ureteral stenosis or renal stenosis and narrow ureteropelvic junction/ureterovesical junction
* Subjects with known impaired renal function from stage IV or known dialysis
* Subjects with chronic hydronephrosis not associated with nephrolithiasis
* Subjects with the following known or suspected diseases: Coagulation disorders, untreated urinary tract infections, renal disease sepsis and marked prostatic hyperplasia
* Subjects with any other disease or condition that, in the opinion of the investigator, could interfere with the purpose of the study (e.g. bleeding that restricts vision in the kidney, problems in the renal tubular system)
* Breastfeeding or pregnant women
* Subjects who may be part of a vulnerable group (e.g. prisoners or developmentally delayed adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Stone free Rate after URS | From enrollment to postoperative follow-up at 2 months.
  To answer the primary research question, a comparison of the SFR between the two surgical procedures is planned using the chi-square test. In order to be able to show a statistically significant difference with regard to the surgical procedures according to the current data situation (75 % vs. 95 %), a sample size of 120 was defined with a power of 80 % and a significance level of 0.025 (the significance correction is made due to the definition of two co-primary endpoints in relation to the definition of freedom from stones).

SECONDARY OUTCOMES:
Surgery Duration | During the procedure
  • Duration of surgery (minutes, continuous): defined as the time from transurethral entry with the cystoscope to ureteral stent insertion in the affected kidney)
Laser duration | during the procedure
  • Laser duration (minutes, continuous): defined as the time until the stone is sufficiently dusted
Basketing duration | during the procedure
  • Basketing duration (minutes, continuous): defined as the time until the fragments are completely captured and removed
Complication | after the procedure up to 1 month
  • Complication rates according to Clavien Dindo (I-IV); the type and number (%) are recorded
Subjective assessment of the operation by the surgeon | During the procedure
  • Subjective assessment of the operation by the surgeon via questionnaire (Likert scales, 1-5): Difficulty 1 (easy) - 5 (very difficult) ,Stone-free 1(no stones) - 5 (2nd look necessary)
Cost | From enrollment to postoperative follow-up at 12 months
  Costs (euros): defined as the costs of hospitalization, surgery, outpatient care and emergency presentation in euros per patient
Frequency of a stone-related event | From enrollment to postoperative follow-up at 3 months.
  Frequency of a stone-related event (defined as an event related to stone treatment, %): Repeat operation: DJ blocked (yes, no), completion of URS in case of residual stone (yes, no), repeat URS in case of stone recurrence (yes, no, side), DJ in case of new stone formation (yes, no, side, type), New stone formation: stone recurrence (yes, no, side), colic (yes, no, side), new imaging (yes, no, type)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Straub, Doctor, Principal Investigator — Technical University of Munich
Locations (1):
- University Hospital rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
The Patient Data is only planned for this Study